CLINICAL TRIAL: NCT07250165
Title: Prospective, Single-arm, Open-label Study of Efficacy and Safety of 532 nm KTP and Microsecond 1064 nm Nd:YAG Laser in Rosacea
Brief Title: Combined Therapy of 532-nm KTP and Microsecond 1064-nm Nd:YAG Laser for Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Yanhong Sun, Attending Physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-2024-0959
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Rosacea
Keywords: Rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined 532 nm KTP + microsecond 1064 nm Nd:YAG laser (Experimental): Participants are allocated to receive combined dual-wavelength laser therapy (microsecond 1064 nm Nd:YAG followed by 532 nm KTP) in a single session, repeated every 3 weeks for a total of three sessions. No anaesthesia is used.
  Interventions: Device: Excel V, Cutera, Brisbane, CA

INTERVENTIONS:
Device: Excel V, Cutera, Brisbane, CA — The facial erythema was treated with 532-nm KTP combined with microsecond 1064-nm ND:YAG laser. Each patient received three consecutive laser treatments with an interval of three weeks . Patients were treated using both laser modules during the same session without anesthesia. Firstly, microsecond 1064-nm Nd:YAG laser (Excel V, Cutera, Brisbane, CA) was applied with an 8 mm spot size, 0.3ms pulse duration, and energy density of 6-7 J/cm². Then, 532-nm KTP laser was used for treatment. When a 10 mm spot size was used, the energy density was 6-9 J/cm² and the pulse duration was 8-15ms; when a 5 mm spot size was used, the energy density was 8-10 J/cm² and the pulse duration was 8-12ms.

SUMMARY:
Rosacea remains a therapeutically challenging, chronic facial dermatosis whose central feature-persistent erythema-often resists topical and systemic agents. In this study we evaluated, for the first time, the simultaneous use of a 532-nm potassium titanyl phosphate (KTP) laser and a microsecond-pulsed 1064-nm Nd:YAG laser as a safe alternative.

DETAILED DESCRIPTION:
Rosacea is an extremely common condition characterised by facial flushing, dilated capillaries and papules and pustules. Both systemic and topical treatments have their drawbacks, such as limited efficacy, intolerable adverse reactions, drug resistance and high recurrence rates. Therefore, it is necessary to explore new treatment methods for rosacea.

Lasers have been used for more than three decades to treat vascular lesions with an excellent safety profile and very low risk of scar formation. Purpura was a common side effect of the previous generation of lasers and has been significantly reduced with the introduction of newer devices. The 532-nm potassium titanyl phosphate (KTP) laser is used for treating vascular cutaneous lesions due to its selective absorption by haemoglobinn, while rarely inducing purpura. However, the 532-nm KTP laser is primarily effective for superficial blood vessels. The long-pulsed 1064-nm neodymium-doped yttrium aluminum garnet (Nd:YAG) laser can penetrate up to 4-6 mm beneath the skin and is effective in treating larger blood vessels. Previous studies have demonstrated that the long-pulsed 1064-nm Nd:YAG laser is effective for both erythematotelangiectatic rosacea (ETR) and papulopustular rosacea (PPR). However, traditional millisecond-domain devices should still be used with caution in darker skin types, and it is associated with an extensive zone of thermal injury and a heightened risk of scar formation. In contrast to millisecond 1064-nm Nd:YAG lasers, microsecond-pulsed lasers deliver energy within the thermal relaxation time of the epidermis, minimizing heat diffusion to surrounding tissues.

Rosacea is a chronic and recurrent dermatologic condition that poses significant therapeutic challenges. While both 532-nm KTP and 1064-nm Nd:YAG lasers demonstrate efficacy in managing rosacea-associated erythema, no single laser system can address all vascular components due to their distinct limitations in penetration depth and vessel selectivity. We need to explore more treatment options. This study aims to evaluate the efficacy and safety of a 532-nm KTP laser combined with a microsecond 1064-nm ND:YAG laser in treating the erythema of rosacea, in order to provide scientific evidence for clinical application.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged between 18 and 65 years, without cognitive impairments, and of any gender
* Patients must meet the 2017 rosacea diagnostic criteria updated by the National Rosacea Society Expert Committee
* The severity of rosacea must be scored at least 2 points on the Clinician's Erythema Assessment (CEA) scale.

Exclusion Criteria:

* if they had undergone any treatments that could influence the prognosis of rosacea within the preceding 8 weeks
* if they had taken photosensitizing or phototoxic medications within the same period
* the presence of other facial conditions that might confound the efficacy assessment
* participation in any drug clinical trial as a subject within the last month
* the presence of severe concurrent diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-08-10 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-02 (Actual)

PRIMARY OUTCOMES:
CEA scores | Baseline to Week 9
  Change from baseline in Clinician Erythema Assessment (CEA) at Week 9; scored 0-4 by blinded photograph review.
CEA success | Baseline to Week 9
  A decrease in CEA of 1 or more is considered as a CEA success

SECONDARY OUTCOMES:
DLQI score | Baseline to Week 9
  The Dermatological Life Quality Index (DLQI) is a validated self-reported questionnaire consisting of 10 questions designed to assess how skin disorders affect a patient's quality of life. The maximum possible score for the DLQI is 30, with higher scores indicating a more significant impact on quality of life.
GAIS score | Week 9
  The global aesthetic improvement scale (GAIS) was used to score the improvement (0 = worse, 1 = unaltered, 2 = improved, 3 = much improved, 4 = very much improved).

OTHER OUTCOMES:
Patient satisfaction | Week 9
  Patient satisfaction was assessed by the patients themselves, with responses categorized as follows: 1 = very satisfied, 2 = satisfied, 3 = neither satisfied nor dissatisfied, 4 = dissatisfied, 5 = very dissatisfied.
Side effects | Baseline to Week 15
  Patients and dermatologists documented any adverse events experienced throughout the study, including pain, heat sensation, erythema, edema, dryness, tightness, itching, purpura, vesicle, hyperpigmentation, hypopigmentation, and scar.

CONTACTS AND LOCATIONS:
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, None Selected, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data (CEA scores, DLQI, GAIS, adverse events) and the study protocol will be made available to qualified researchers beginning 6 months after primary publication. Proposals must be approved by the corresponding author and institution; data will be shared via secure file transfer with a signed data-use agreement.